CLINICAL TRIAL: NCT06429111
Title: Effectiveness and Safety in Maternal and Neonatal Outcomes of Waterbirth Compared to Delivery in Women Using Epidural Analgesia
Brief Title: Effectiveness and Safety in Maternal and Neonatal Outcomes in Water Birth.
Status: Completed | Type: Observational
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Collaborators: Universitat Jaume I (Other); Hospital Universitario de la Plana (Other)
Responsible Party: Principal Investigator, Soledad Carregui Villar, Principal Investigator, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Other Study IDs: water birth
Record Dates: First submitted 2024-05-15; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Natural Childbirth; Water Birth; Neonatal Asphyxia; Outcome, Adverse Birth; Labor Pain; Obstetric Pain
MeSH Terms: conditions — Asphyxia Neonatorum; Pregnancy Complications; Labor Pain | interventions — Analgesia, Epidural

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- low-risk pregnant women who freely chooses to use epidural analgesia during labor: * Pregnant women at term with normal pregnancy without the presence of maternal and neonatal risk factors who meet criteria according to the protocol for the use of water and who choose epidural analgesia at the time of admission to the dilatation room in active labor.
  * Over 17 years of age
  * Psychic and cognitive capacity for decision making
  * Willingness to take part in the study and signature of the informed consent form.
  * Absence of ideomatic barrier
  Interventions: Procedure: Epidural analgesia
- low-risk pregnant woman who freely chooses the use of water during childbirt: Pregnant women at term with normal pregnancy without the presence of maternal and neonatal risk factors who meet criteria according to the protocol for the use of water and who choose immersion water at the time of admission to the dilatation room in active labor.
  * Over 17 years of age
  * Psychic and cognitive capacity for decision making
  * Willingness to take part in the study and signature of the informed consent form.
  * Absence of ideomatic barrier
  Interventions: Procedure: Immersion water

INTERVENTIONS:
Procedure: Epidural analgesia — Consists of a central nerve block by injecting a local anesthetic near the nerves that transmit pain, in the lumbar region, for pain relief during labor.
  Groups: low-risk pregnant women who freely chooses to use epidural analgesia during labor
Procedure: Immersion water — Consists of the use of hot water immersion in a birthing tub during labor and/or delivery.
  Groups: low-risk pregnant woman who freely chooses the use of water during childbirt

SUMMARY:
Childbirth is a unique and non-transferable experience in the life of a woman, her partner and her family. It is a very intense process that requires accompaniment and, in the vast majority of cases, requires analgesic support in order to overcome this life event in an optimal and atraumatic way.

Among the analgesic methods for pain relief during the labor process, there are pharmacological and non-pharmacological methods. From the evidence we know that the most effective pharmacological method is epidural analgesia (EA), while the most recognized non-pharmacological method is immersion in hot water (bathtub) for dilatation and delivery, called waterbirth(WB) At present there is controversy and doubts about the increase in the number of interventions involving the use of epidural analgesia, but there is also controversy about the safety of the use of water, especially in those processes where the birth ends in water. Given the popularity of these two methods, the aim is to study and compare the maternal and neonatal outcomes derived from the use of both methods in order to provide greater knowledge to women in their decision making.

DETAILED DESCRIPTION:
At present there is controversy and doubts about the increase in the number of interventions involving the use of epidural analgesia(EA), but there is also controversy about the safety of the use of water, especially in those processes where the birth ends in water, called Waterbirth (WB). Given the popularity of these two methods, the aim is to study and compare the maternal and neonatal outcomes derived from the use of both methods in order to provide greater knowledge to women in their decision making.

For this purpose, a prospective observational study will be carried out in low-risk pregnant women (who do not present any complication at the time of delivery) who freely choose one or the other method at the beginning of their labor process. For this reason, the socio-demographic characteristics, the obstetric interventions carried out during the process, the results, the possible maternal and neonatal complications, aspects of breastfeeding, as well as the evaluation of the degree of satisfaction will be described and compared between the two groups.

The study was carried out at the Hospital Universitario La Plana, a referral center for normal childbirth, where the healthcare team has experience in the management of both methods. After obtaining the approval of the ethics committee (CEI), recruitment of the cases began and was carried out between June 2020 and February 2023. Overall, 642 cases were recruited, distributed in a total of 359 women who chose water immersion, of whom 40 women subsequently opted for epidural analgesia and 283 women who chose epidural analgesia initially. Women who completed the water birth totaled 263 cases.

The data concerning clinical variables were extracted from the electronic clinical records of the medical history of both the mother and the neonate and subsequently transcribed into a web portal designed to facilitate the transcription of the multiple variables. The final database is exploited from this web portal in Excel format and exported to the Statistical Package for Social Sciences (SPPSS) program version for subsequent analysis.

The variables collected for subsequent analysis are classified into sociodemographic variables, maternal clinical variables, neonatal clinical variables and satisfaction variables.

Satisfaction will be measured according to the Women's Satisfaction with Childbirth Experience Scale. Translated and validated version of the Mackey Satisfaction Childbirth Rating Scale. This scale, originally developed in English, measures women's satisfaction with the experience of childbirth and childbirth. It is a self-completed questionnaire, which is administered to the woman before discharge from the hospital. It consists of 34 items grouped into five subscales referring to the woman (9 items), the partner (2 items), the newborn (3 items), the midwife (9 items) and the obstetrician (8 items). It also contains a subscale for overall assessment of the experience (3 items). Each item is evaluated on a 5-point Likert scale ranging from very dissatisfied (1) to very satisfied (5), with a neutral central value. The final score of the scale is obtained by adding the values assigned to each item, so that the higher the score, the greater the satisfaction. Similarly, partial scores can be obtained for each subscale.

In our study, the obstetrician dimension was eliminated since in women in the waterbirth group the care offered during the process is carried out by the midwife and the women do not receive assistance from the physician.

OBJECTIVES

The General Objective of the study is to compare the effectiveness and safety of the use of water during dilatation and delivery versus the administration of epidural analgesia in low-risk women.

The Specific Objectives are:

. To describe and compare between the two groups the socio-demographic and obstetric characteristics of the pregnant women participating in the study (age, parity, weeks of gestation, type of breastfeeding chosen, level of education, country of origin, vagino-rectal colonization by beta-hemolytic streptococcus, weight of the NB, sex).

To describe and compare between the two groups the difference in obstetric interventions (administration of oxytocin, amniorrhexis, bladder catheterization, fetal calcium levels, need for other analgesic support during the process, episiotomy and position adopted by the mother for the birth).

* To describe and compare between both groups the maternal outcomes of the process (end of labor, dilatation time, expulsion time, perineal tears, duration of admission, visits to the emergency department during the first month of life).
* To describe and compare between both groups the possible maternal complications that occur in the process (instrumental delivery, cesarean section, Fetal Healt rate(FHR),alterations, III and IV degree tear, presence of obstetric emergency, intrapartum fever and puerperal infection).
* To describe and compare between both groups the neonatal outcomes (Apgar of the newborn at one minute, 5 and 10 minutes, cord arterial pH, venous arterial pH, base excess, need for neonatal ventilation support, admission to the neonatal unit or Neonatal Intensive care unit (NICU), reason and duration of admission).
* To describe and compare between both groups the initiation and evolution of breastfeeding (initial choice, breastfeeding at discharge, neonatal alertness at birth, type of latch, supplementation during hospital stay).
* To describe and compare between the two groups the degree of satisfaction with childbirth between the epidural and water use groups according to the validated Mackey Scale, assessing the dimensions of woman, partner, newborn, midwife and overall assessment of the experience.

TREATMENT OF SUBJECTS - SAMPLING TECHNIQUE

The non-probabilistic consecutive sampling technique will be used, offering the study to women who meet the inclusion criteria and have no exclusion criteria.

The women will be recruited in the Delivery Service when the pregnant woman finishes the delivery process, while still in the dilation room, and who meet the inclusion criteria and have no exclusion criteria. After the information, the patient will be offered an information sheet and the informed consent form to be signed before leaving the delivery room. The variable recorded in the form of the labor dilatation sheet of the mother's medical history that defines whether the woman is low risk at the time of delivery will be taken into account, this characteristic is defined in the partogram and is a mandatory field that is filled in by the professional to the question "candidate use of water" YES/NO to alert the researcher about the possible case to be considered in the study, this response is conditioned by the protocol for the use of water available at the Hospital de La Plana (the characteristics that indicate whether or not the use of water in childbirth is indicated are clearly defined). After delivery, the midwife will offer the woman the possibility of entering the study, offering her the information sheet and the informed consent form that she will have to sign before discharge from the hospital. In the event that the consent and information is not offered in the delivery service for any reason, it can be done later as long as it is before discharge from the hospital.

Entry into the study will not influence routine clinical practice, since it does not involve any action on the subjects under study. The intervention will be in the analysis of the variables to be studied, this implies the consent of the woman for the exploitation of the data from her Electronic Medical Record and that of her newborn through the forms that are usually used in all childbirth processes. On the other hand, it is necessary to fill in a satisfaction questionnaire, which will be given by the midwife before the woman leaves the delivery service. This questionnaire can be completed from the postpartum period until the woman is discharged from the hospital, and will be collected by the midwife who visits the hospital ward during the days that the woman remains hospitalized, before discharge.

. Before starting the study, a meeting will be held to review the protocol, the data collection booklet and the guidelines to be followed by the personnel involved in the study.

The researcher is committed to compliance with the Organic Law 3/2018, of December 5, on Personal Data Protection (LOPD) and guarantee of digital rights, published in the Boletin Oficial del Estado (BOE), as wel as Regulation (EU) 2016/679 of the European Parliament. The data collected for the study will be pseudonymized, so that it does not include information that can identify patients.

In accordance with Law 41/2002, of November 14, 2002, basic law regulating patient autonomy and rights and obligations regarding information and clinical documentation, all potential candidates will be given an informative document of the study and informed consent so that they can make a rational, free decision in accordance with their values and preferences. No patient can be included in the study without prior informed consent.

The investigator consents, when signing the protocol, to adhere to the instructions and procedures described in them and thus follow the principles of good clinical practice that they imply.

The investigator submitted the relevant documentation to the Research and Ethics Committee (CEI). The study was not initiated until CEI approval was obtained.

Similarly, the managers and the management team were informed for their express consent.

The safety of the study will be controlled through the delivery staff of the Hospital Universitario La Plana, since this study not modify the usual clinical practice by not performing any intervention required by the study in any of the groups.

In the design of the study, priority is given to not randomizing the sample, since ethically, the woman's ability to choose and the fulfillment of her expectations regarding childbirth are prioritized.

The researcher attaches a declaration of absence of conflict of interest. This study will be carried out according to the Standards of Good Clinical Practice and in accordance with the Declaration of Helsinki 1975, amended in 1983. Patients' names and initials will not be included.

DATA MANAGEMENT AND ARCHIVING OF RECORDS

The data necessary for carrying out the study will be collected from the Pregnancy Chart, which classifies whether the pregnant woman has any risk factors, from the hospital medical record entered in the Conficita program of the Hospital Universitario La Plana, where we will access the Obstetric Admission Sheet, the Dilatation-Delivery Sheet, the Newborn Sheet and the Neonatal Follow-Up Sheet in order to collect the variables described in the study. These variables will be collected in a Data Collection Notebook (Annex II).

Subsequently, these data will be collected in the SPSS database and stored in a Clinical Research File (FIC), included in the FIC of the research project of the Department of Health of the Hospital La Pana, attached to the FIC whose owner is the Conselleria de Sanitat. Only the researchers will have access to these data; their sole purpose will be to carry out the present study and the data analysis will be performed with the help of the SPSS statistical package for Windows.

On the occasion of the study, a file will be generated with all the documentation of the study, which will be kept by the researcher. The study documentation will be kept for the time required by current legislation, after which it will be destroyed according to the rules of the service on destruction of documents with personal information.

The investigator allows direct access to the data or source documents for monitoring, auditing and review by the IRB. The study may be audited by the Health Authorities during the study or even when the study is completed, to assess compliance with Good Clinical Practice guidelines.

No data revealing the identity of the patients should leave the center.

PUBLICATION POLICY

The results of the study will be the property of the investigator who will establish the publication policy. In addition, the anonymity of the patients participating in the study will be guaranteed at all times.

This work is a doctoral thesis of the Biomedical Sciences program of the Universitat Jaume I of Castellón, tutored by Dr. Eladio Collado Boira, Dr. Eva Moya Artuñedo and Dr. Ricardo Tosca Segura.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at term with normal pregnancy without the presence of maternal and neonatal risk factors that preclude the use of water and epidural analgesia at the time of admission to the delivery room.

Pregnant women who are 18 years of age or older or who will turn 18 in the year of delivery.

* Have the psychic and cognitive capacity to make decisions.
* Desire to be part of the study and signature of informed consent to participate in the study.

Exclusion Criteria:

* .Presence of any maternal or fetal risk factor that precludes the choice of water or epidural analgesia at the time of admission to the dilation room in active labor.

Under 17 years of age or under 18 years of age in the year of delivery.

.Ideomatic barrier that makes it impossible for the patient to understand the study and to agree to the informed consent, .Unwillingness to participate or failure to sign the informed consent form.

Ages: 17 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The Hospital Universitario La Plana is the reference center of the Health Department No. 3, is a regional hospital located in the city of Vila-real, province of Castellon.
  Candidates for participation in the study are full-term pregnant women who meet the inclusion criteria and who are admitted to the dilation room during the active labor period in the Delivery Service of the Hospital Universitario La Plana during the period from April 2020 to June 2023.
Sampling Method: Non-Probability Sample
Enrollment: 642 (Actual)
Dates: Start 2020-06-06 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Completion of labor | 24 hours
  How labor is terminated :
  Normal in water Normal underwater Instrumented delivery Cesarean section
intrapartum administration of oxytocin | 24 hours
  Yes/no intrapartum oxytocin required
Amniotomy | 24 hours
  If intrapartum amniotomy is needed YES/NO
presence of fetal heart rate abnormalities Frequency of non-reassuring or pathological episodes in the cardiotocographic recording. | 24 hours
  Frequency of non-reassuring or pathological episodes in the cardiotocographic recording.
  (Scale)
Number of bladder catheterizations | Up to 24 hours
  Number of times bladder catheterization is performed during the delivery process (Scale)
Number of scalp blood determinations | Up to 24 hours
  Determination of pH and lactate from fetal scalp blood to study the management of intrapartum fetal hypoxia. Only when when there is suspicion of risk of loss of fetal well-being due to a non-reassuring or pathological cardiotocographic monitor.
  (Scale)
Intrapartum fever | Up tu 24 hours
  Presence of intrapartum fever YES/NO
Presence of obstetric emergency | Up to 24 hours
  An obstetric emergency is considered to be the occurrence of any episode of:
  Cord rupture puerperal hemorrhage Shoulder impaction Manual removal of placenta Risk of loss of fetal well-being (Nominal)
Perineal tear | Up to 24 hours
  Injury to the genital tract due to spontaneous trauma as a result of childbirth. These traumas are classified according to Sultan 1999 according to the injury produced:
  First degree: Injury to the perineal skin and mucosa. Second degree: Injury to perineal muscles without affecting the anal sphincter. Third degree a.- Injury that reaches the external anal sphincter affecting less than 50%.
  Third degree b.- Injury reaching the external anal sphincter affecting more than 50%.
  Third degree c.- Injury reaching the complete external anal sphincter and internal anal sphincter.
  Fourth degree: Injury to the external anal sphincter plus the internal anal sphincter plus the anal epithelium.
  (Nominal)
Apgar score at one minuto of life of the neonate. | Up to 24 hours
  A one-minute assessment of five items that determine a numerical value called the "Apgar test" that evaluates cardiac activity, respiratory effort, reflexes, muscle tone and skin color.
  If the value is less than or equal to 7, it is interpreted as a poor neonatal adaptation; if it is greater than 7, it is interpreted as an adequate adaptation.
  (Scale)
Apgar score at five minuts of life of the neonate. | Up to 24 hours
  A five minutes assessment of five items that determine a numerical value called the "Apgar test" that evaluates cardiac activity, respiratory effort, reflexes, muscle tone and skin color.
  If the value is less than or equal to 7, it is interpreted as a poor neonatal adaptation; if it is greater than 7, it is interpreted as an adequate adaptation.
  (Scale)
Arterial cord blood ph | Up to 24 hours
  Value determining the analysis of blood samples from the umbilical cord artery after birth. The purpose of this analysis is to determine the degree of possible fetal hypoxia suffered by the newborn during delivery. The blood sample will be taken without clamping the umbilical cord in the case of late cord. A value lower than 7.10 can be interpreted as a higher risk of fetal hypoxia.
  (Scale)
Neonatal ventilation support | Up to 24 hours
  If the neonate requires after birth support with positive ventilation, oxygen administration or intubation. YES/NO
Presence of distress neonatal | Up to 48 hours
  Presence of respiratory distress in the neonate during the first two hours of life.
  YES/NO
Neonatal admission | Up to 30 days
  Describes if the neonate needs to be admitted to the neonatal unit. YES/NO
Neonatal sepsis | Up to 30 days
  Describes whether neonatal sepsis has occurred.YES/NO
Presence of hypoxic ischemic encephalopathy | 1 month
  Describes whether the neonate has a diagnosis of hypoxic ischemic encephalopathy.
Maternal infection | Up to 1 month
  Presence of any type of maternal infection in the postpartum period (urinary tract infection, endometritis, mastitis or others), YES/NO
Breastfeeding upon hospital discharge | Up to 1 week
  Type of breastfeeding established at hospital discharge:
  Breastfeeding Artificial breastfeeding Mixed breastfeeding
Visits to the hospital emergency department during the first month postpartum | Up to1 month
  Number of urgent hospital visits made by the woman during the first postpartum month.
  (Scale)
Maternal satisfaction | Up to 3 days
  Measured according to the validation of the Mackey Childbirth Satisfaction Rating Scale. It consists of 34 items grouped in five subscales referring to the woman (9 items), the partner (2 items), the newborn (3 items), the midwife (9 items) and the obstetrician (8 items). It also contains a subscale for overall assessment of the experience (3 items). Each item is evaluated on a 5-point Likert scale ranging from very dissatisfied (1) to very satisfied (5), with a neutral central value. The final score of the scale is obtained by adding the values assigned to each item, so that the higher the score, the greater the satisfaction. Similarly, partial scores can be obtained for each subscale.
  The questionnaire is offered to the woman in the postpartum period and is collected before discharge from the hospital.

SECONDARY OUTCOMES:
cervical dilatation at the time of choice of analgesic method | Up to 24 hours
  cervical dilatation in centimeters at the time of analgesic method choice
group b streptococcus colonization during gestation | Up to 24 hours
  vagino-rectal colonization with positive result for group B streptococcus at the time of delivery
Duration of the dilatation phase | Up to 24 hours
  Duration in minutes of the dilation phase from admission to the delivery room until the beginning of the active expulsion period (Scale)
Duration of the active second stage of labor | Up to 24 hours
  Duration in minutes of the active phase of the second stage of labor from the start of pushing to delivery.
Type of expulsion | Up to 24 hours
  Type of pushes performed by the woman during the second stage of labor. They can be directed pushes or spontaneous pushes.
Management of the third stage of labor | Up to 24 hours
  Management of third stage of labor:
  * Active if oxytocin and directed labor are used
  * Passive -physiologic management
newborn birth weight | Up to 24 hours
  newborn birth weight expressed in grams
sex of the newborn | Up to 24 hours
  sex of the newborn
  * male
  * female
Breastfeeding chosen after birth | Up to 24 hours
  Breastfeeding chosen after birth
  * Breastfeeding
  * Artificial feeding
Type of latch-on of the baby at the onset of breastfeeding during the first two hours postpartum | Up to 48 hours
  * Spontaneous onset
  * Spontaneous onset
  * Onset with maternal support
  * Onset with professional help
  * No initiation
Reason for admission | Up to 1 month
  * Infectious risk
  * Glycemic control
  * Jaundice
  * Feeding problems
  * Fetal malformations
  * Distress
  * Neonatal Sepsis
  * Transfer to neonatal ICU
  * Other
  * No admission
Supplementation during hospital stay | At the time of hospital discharge
  Number of times the baby is offered supplementation with formula during hospital stay (Scale)
Length of stay in days | At the time of hospital discharge
  Days the newborn stays in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Soledad Carregui Vilar, Midwife, Principal Investigator — Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Locations (1):
- Hospital Universitario La Plana, Vila-real, Castellon, Spain

IPD SHARING:
Plan to Share IPD: Undecided
We plan to publish the data available to other researchers, including the study protocol, the protocol for water use at la plana university hospital and the informed consent form.

REFERENCES:
- [Background] Cluett ER, Burns E, Cuthbert A. Immersion in water during labour and birth. Cochrane Database Syst Rev. 2018 May 16;5(5):CD000111. doi: 10.1002/14651858.CD000111.pub4. PMID 29768662
- [Background] Anim-Somuah M, Smyth RM, Cyna AM, Cuthbert A. Epidural versus non-epidural or no analgesia for pain management in labour. Cochrane Database Syst Rev. 2018 May 21;5(5):CD000331. doi: 10.1002/14651858.CD000331.pub4. PMID 29781504
- [Background] Shaw-Battista J. Systematic Review of Hydrotherapy Research: Does a Warm Bath in Labor Promote Normal Physiologic Childbirth? J Perinat Neonatal Nurs. 2017 Oct/Dec;31(4):303-316. doi: 10.1097/JPN.0000000000000260. PMID 28520654
- [Background] Lewis L, Hauck YL, Butt J, Hornbuckle J. Obstetric and neonatal outcomes for women intending to use immersion in water for labour and birth in Western Australia (2015-2016): A retrospective audit of clinical outcomes. Aust N Z J Obstet Gynaecol. 2018 Oct;58(5):539-547. doi: 10.1111/ajo.12758. Epub 2018 Jan 17. PMID 29344940
- [Background] Bovbjerg ML, Cheyney M, Caughey AB. Maternal and neonatal outcomes following waterbirth: a cohort study of 17 530 waterbirths and 17 530 propensity score-matched land births. BJOG. 2022 May;129(6):950-958. doi: 10.1111/1471-0528.17009. Epub 2021 Dec 1. PMID 34773367
- [Background] Liu Y, Liu Y, Huang X, Du C, Peng J, Huang P, Zhang J. A comparison of maternal and neonatal outcomes between water immersion during labor and conventional labor and delivery. BMC Pregnancy Childbirth. 2014 May 6;14:160. doi: 10.1186/1471-2393-14-160. PMID 24886438
- [Background] Yu M, Qian H, Gan M. Comparison of different interventions for the reduction of labor pain: A systematic review and network meta-analysis. Medicine (Baltimore). 2024 Mar 8;103(10):e37047. doi: 10.1097/MD.0000000000037047. PMID 38457589
- [Background] McKinney JA, Vilchez G, Jowers A, Atchoo A, Lin L, Kaunitz AM, Lewis KE, Sanchez-Ramos L. Water birth: a systematic review and meta-analysis of maternal and neonatal outcomes. Am J Obstet Gynecol. 2024 Mar;230(3S):S961-S979.e33. doi: 10.1016/j.ajog.2023.08.034. Epub 2024 Jan 9. PMID 38462266
- [Background] Seed E, Kearney L, Weaver E, Ryan EG, Nugent R. A prospective cohort study comparing neonatal outcomes of waterbirth and land birth in an Australian tertiary maternity unit. Aust N Z J Obstet Gynaecol. 2023 Feb;63(1):59-65. doi: 10.1111/ajo.13555. Epub 2022 Jul 7. PMID 35796252
- [Background] Zhang G, Yang Q. Comparative Efficacy of Water and Conventional Delivery during Labour: A Systematic Review and Meta-Analysis. J Healthc Eng. 2022 Mar 29;2022:7429207. doi: 10.1155/2022/7429207. eCollection 2022. PMID 35392147
- [Background] Ulfsdottir H, Saltvedt S, Edqvist M, Georgsson S. Management of the active second stage of labor in waterbirths compared with conventional births - a prospective cohort study. Midwifery. 2022 Apr;107:103283. doi: 10.1016/j.midw.2022.103283. Epub 2022 Feb 8. PMID 35172265
- [Background] Reviriego-Rodrigo E, Ibargoyen-Roteta N, Carregui-Vilar S, Mediavilla-Serrano L, Uceira-Rey S, Iglesias-Casas S, Martin-Casado A, Toledo-Chavarri A, Ares-Mateos G, Montero-Carcaboso S, Castello-Zamora B, Burgos-Alonso N, Moreno-Rodriguez A, Hernandez-Tejada N, Koetsenruyter C. Experiences of water immersion during childbirth: a qualitative thematic synthesis. BMC Pregnancy Childbirth. 2023 May 29;23(1):395. doi: 10.1186/s12884-023-05690-7. PMID 37248449
- [Background] Burns E, Feeley C, Hall PJ, Vanderlaan J. Systematic review and meta-analysis to examine intrapartum interventions, and maternal and neonatal outcomes following immersion in water during labour and waterbirth. BMJ Open. 2022 Jul 5;12(7):e056517. doi: 10.1136/bmjopen-2021-056517. PMID 35790327
- [Background] Vanderlaan J, Hall P. Systematic Review of Case Reports of Poor Neonatal Outcomes With Water Immersion During Labor and Birth. J Perinat Neonatal Nurs. 2020 Oct/Dec;34(4):311-323. doi: 10.1097/JPN.0000000000000515. PMID 33079805
- [Background] Ulfsdottir H, Saltvedt S, Georgsson S. Women's experiences of waterbirth compared with conventional uncomplicated births. Midwifery. 2019 Dec;79:102547. doi: 10.1016/j.midw.2019.102547. Epub 2019 Sep 30. PMID 31610362
- [Background] Committee Opinion No. 679 Summary: Immersion in Water During Labor and Delivery. Obstet Gynecol. 2016 Nov;128(5):1198-1199. doi: 10.1097/AOG.0000000000001765. PMID 27776069